CLINICAL TRIAL: NCT02141503
Title: Clinical Biomarkers in Alpha-Mannosidosis
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140106; 14-CH-0106
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-11-29

CONDITIONS: Alpha-Mannosidosis
Keywords: Biomarkers; Alpha-Manosidosis
MeSH Terms: conditions — alpha-Mannosidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

SUMMARY:
Background:

- Alpha-mannosidosis is a rare inherited disorder. It causes problems in many organs and tissues of the body. It can occur in children and adults. Because there is no treatment for this disease, researchers want to find out more about it.

Objective:

- To learn more about Alpha-mannosidosis.

Eligibility:

- People ages 5-60 with Alpha-mannosidosis.

Design:

* Participants will be recruited from patient support organizations and medical genetics clinics.
* Participants will have 3 study visits, about once a year. A final evaluation will be made after 3 years.
* Participants will have a medical history and a physical exam.
* Blood samples and a urine sample will be collected.
* Cerebrospinal fluid will be collected. A small area of the lower back will be numbed with medicine. A thin needle will be inserted between the spine bones. About 2 tablespoons of spinal fluid will be removed.
* Brain magnetic resonance spectroscopy (MRS) scans will be done at each visit. MRS uses a strong magnetic field and radio waves to take pictures of chemicals in the brain with a scanner. The participant will lie on a table that can slide in and out of the cylinder. While in the scanner the participant will hear loud knocking noises. They will get earplugs or earmuffs to muffle the sound. Medicines might be used to keep the participant asleep during the MRS.
* Participants will have a skin biopsy at the first visit only. A small area of the participant s skin will be numbed. A small circle of skin will be removed with a biopsy tool.

DETAILED DESCRIPTION:
Alpha-mannosidosis (AMD) is an inherited lysosomal storage disorder caused by mutations in the LAMAN gene, which encodes lysosomal alpha-mannosidase and is characterized by neurodevelopmental delay, mild immune deficiency, facial and skeletal abnormalities, hearing impairment, intellectual disability, muscle weakness and ataxia. The progression of neuromuscular and skeletal deterioration is insidious, occurring over several decades, rendering most patients wheel-chair dependent. No consistently successful treatment is available. To better characterize the biochemical phenotype and natural history of this disorder, we will study 15 patients with AMD, ranging in age from five to 60 years, recruited from Departments of Biochemical Genetics and Medical Genetics at university medical centers mainly in the US and Canada or referred by the Intl Society for Mannosidosis & Related Diseases. Participants in the study will visit the NIH Clinical Center 2-3 days on an outpatient basis and will undergo clinical and biochemical evaluations to establish reliable clinical

benchmarks and to identify cerebrospinal fluid biomarkers that could serve as candidate

surrogate markers of treatment effect in future clinical trials. The protocol will take advantage of the NICHD Biomedical Mass Spectrometry Facility to generate CSF proteomic profiles. Patients will also undergo MR spectroscopy (under sedation/anesthesia, if appropriate) in order to establish the phenotypic baseline and for possible utility as a guide for natural history and/or treatment outcomes in future studies. If the pre-clinical components of this proposal prove promising, the prospect of a recombinant adeno-associated viral gene therapy trial involving a brain-directed (intrathecal) approach for AMD would be possible within 3 years.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Must have a verifiable diagnosis of AMD based on clinical, biochemical and/or molecular grounds, including increased urinary excretion of mannose-rich oligosaccharides, decreased acidic -mannosidase activity in leukocytes or other nucleated cells, and/or mutations in two alleles of the LAMAN gene.
  2. Must be at least five years old.

EXCLUSION CRITERIA:

1. Significant systemic or major disease including congestive heart failure, coronary artery disease, cerebrovascular disease and pre-existing or recent onset pulmonary disease, renal failure, organ transplantation, decompensated liver disease, serious psychiatric disease, or malignancy that in the opinion of the investigator would preclude successful participation..
2. Pregnancy. We will perform a urine pregnancy test on all post-menarcheal female subjects on the same day as the history and physical exam, prior to MRI. If pregnancy is identified, we will follow Maryland state law in place at the time concerning parental notification. In the event a woman becomes pregnant during the study, she will be withdrawn from all study procedures, but the study team will follow up with the participant regarding the pregnancy outcome.

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2014-07-24; Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Identify cerebrospinal fluid biomarkers that could serve as candidate surrogate markers of treatment effect in a future clinical trial. | Baseline
  Identify cerebrospinal fluid biomarkers that could serve as candidate surrogate markers of treatment effect in a future clinical trial.

SECONDARY OUTCOMES:
Establish reliable clinical benchmarks for alpha-mannosidosis. | Ongoing
  Establish reliable clinical benchmarks for alpha-mannosidosis.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen G Kaler, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Malm D, Nilssen O. Alpha-mannosidosis. Orphanet J Rare Dis. 2008 Jul 23;3:21. doi: 10.1186/1750-1172-3-21. PMID 18651971
- [Background] Schutzer SE, Liu T, Natelson BH, Angel TE, Schepmoes AA, Purvine SO, Hixson KK, Lipton MS, Camp DG, Coyle PK, Smith RD, Bergquist J. Establishing the proteome of normal human cerebrospinal fluid. PLoS One. 2010 Jun 11;5(6):e10980. doi: 10.1371/journal.pone.0010980. PMID 20552007
- [Background] Magnitsky S, Vite CH, Delikatny EJ, Pickup S, Wehrli S, Wolfe JH, Poptani H. Magnetic resonance spectroscopy of the occipital cortex and the cerebellar vermis distinguishes individual cats affected with alpha-mannosidosis from normal cats. NMR Biomed. 2010 Jan;23(1):74-9. doi: 10.1002/nbm.1430. PMID 19743435